CLINICAL TRIAL: NCT05092269
Title: A Phase 3, Multicenter, Open-label, Basket, Long-term Extension Study of Ustekinumab in Pediatric Clinical Study Participants (2 to <18 Years of Age)
Brief Title: A Long-term Extension Study of Ustekinumab in Pediatric Participants
Acronym: UNITED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR109074; CNTO1275ISD3001 (Other: Janssen Research & Development, LLC); 2020-004457-76 (EudraCT Number); 2022-501067-40-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease; Colitis, Ulcerative; Arthritis, Psoriatic
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Arthritis, Psoriatic | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ustekinumab (Experimental): Participants will have continued access to ustekinumab for primary study (CNTO1275CRD1001, CNTO1275PUC3001, CNTO1275CRD3004, CNTO1275JPA3001) participants who in the opinion of the investigator will continue to benefit from ustekinumab therapy. All blinded participants who enroll in the long-term extension (LTE) from blinded primary studies with both every 8 weeks (q8w) and every 12 weeks (q12w) dosing groups just prior to the end of the primary study will be assigned to the q8w dosing regimen. Participants enrolling in the LTE from an unblinded primary study will remain on the final dosing regimen that they were receiving in the primary study. Participants enrolling from the Exposure Optimization Substudy may be eligible to remain on the every 4 weeks (q4w) dosing regimen.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Ustekinumab will be administered as a SC injection.
  Other Names: STELARA

SUMMARY:
The purpose of this study is to collect long-term safety data of subcutaneous (SC) ustekinumab

ELIGIBILITY:
Inclusion Criteria:

* Must have completed the dosing planned in the primary pediatric ustekinumab study
* Benefit of continued ustekinumab therapy (that is, a clinical response or clinical remission as defined in the primary study at the final efficacy visit of the primary study)
* Parent(s) (preferably both if available or as per local requirements), legal guardian(s) or their legally acceptable representative must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to allow the child to participate in the study. Assent is also required of children capable of understanding the nature of the study (typically 7 years of age and older) as described in Informed Consent Process. An adolescent who signs the assent form will be given the opportunity to sign an adult ICF at a later visit when they reach the age of majority during the study to indicate that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Must be willing and able to adhere to the lifestyle restrictions specified in this protocol
* Females of childbearing potential must have a negative urine pregnancy test at enrollment and prior to study intervention administration

Exclusion Criteria:

* Are pregnant, nursing, or planning pregnancy or fathering a child
* Have had any of (a) confirmed severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2 [COVID-19]) infection (test positive), or (b) suspected SARS-CoV-2 infection (clinical features without documented test results), or (c) close contact with a person with known or suspected SARS-CoV-2 infection: Exception: (i) may be included with a documented negative result for a validated SARS-CoV-2 test: obtained at least 2 weeks after conditions (a), (b), (c) above (timed from resolution of key clinical features if present, example, fever, cough, dyspnea) and (ii) with absence of all conditions (a), (b), (c) above during the period between the negative test result and the baseline study visit
* Taken any disallowed therapies as noted in the primary study, before the planned first long-term extension (LTE) dose of study intervention
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participants who receive a live vaccination may be permitted to remain in the study, if approved by the sponsor and study intervention is held for a period of time specified by the sponsor. Receipt of a live severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) vaccine (against the virus that causes Coronavirus Disease 2019 [COVID-19]) is not automatically an exclusion criterion and must be discussed with the medical monitor

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 6 years and 4 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Number of Participants With Serious Adverse Events (SAEs) | Up to 6 years and 4 months
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants with AEs Leading to Discontinuation of Study Intervention | Up to 6 years and 4 months
  Number of participants with AEs leading to discontinuation of study intervention will be reported.
Number of Participants with AEs of Interest | Up to 6 years and 4 months
  Number of participants with AEs of special interest (any newly identified malignancy case of active tuberculosis [TB], or opportunistic infection occurring after the first administration of study intervention[s]) will be reported.
Number of Participants with Abnormalities in Clinical Laboratory Parameters | Up to 6 years and 4 months
  Number of participants with abnormalities in clinical laboratory parameters (such as hematology and serum chemistry) will be reported.
Number of Participants with Injection-site Reactions | Up to 6 years and 4 months
  Number of participants with injection-site reactions will be reported. An injection-site reaction is any adverse reaction at a subcutaneous (SC) study intervention injection-site.
Number of Participants With AEs of Worsening of the Disease | Up to 6 years and 4 months
  Number of participants with AEs of worsening of the disease will be reported.
Number of Participants With Concomitant Therapy due to Loss of Response | Up to 6 years and 4 months
  Number of participants with concomitant therapy due to loss of response will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (47):
- United States (4):
  - Children's Center For Digestive Healthcare, Llc, Atlanta, Georgia
  - Mount Sinai, New York, New York
  - Levine Childrens at Atrium Health, Charlotte, North Carolina
  - Pediatric Specialists Of Virginia, Fairfax, Virginia
- Argentina (3):
  - STAT Research S A, Buenos Aires
  - Hospital de Ninos de Cordoba, Córdoba
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Belgium (5):
  - Huderf, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Gent, Ghent
  - UZ Brussel, Jette
  - Uz Gasthuisberg, Leuven
- Hôpital Necker, Paris, France
- Germany (2):
  - Universitaetsklinikum der RWTH Aachen, Aachen
  - Charite Universitatsmedizin Berlin Campus Virchow Klinikum, Berlin
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Borsod Abauj Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Szabolcs Szatmar Bereg Varmegyei Oktatokorhaz, Nyíregyháza
  - Szegedi Tudomanyegyetem, Szeged
- Israel (3):
  - Yitzhak Shamir Medical Center, Beer Yaakov
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Fondazione IRCCS Ca Granda Ospedale Policlinico Di Milano, Milan, Italy
- Japan (8):
  - Juntendo University Hospital, Bunkyō City
  - Gunma University Hospital, Gunma
  - Kindai University Nara Hospital, Ikoma
  - Kurume University Hospital, Kurume
  - Saitama Childrens Medical Center, Saitama Shi
  - Miyagi Children's Hospital, Sendai
  - National Center for Child Health and Development, Setagaya Ku
  - Mie University Hospital, Tsu
- Poland (6):
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Korczowski Bartosz Gabinet Lekarski, Rzeszów
  - Centrum Zdrowia Dziecka i Rodziny im Jana Pawla II w Sosnowcu Sp z o o, Sosnowiec
  - GASTROMED Sp. z o.o., Torun
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
  - Medical Network, Warsaw
- Hosp. Univ. I Politecni La Fe, Valencia, Spain
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Ankara
  - Cerrahpasa Medical Faculty Hospital, Istanbul
- United Kingdom (6):
  - Birmingham Children's Hospital, Birmingham
  - Addenbrookes Hospital, Cambridge
  - Royal London Hospital, London
  - Great Ormond Street Hospital, London
  - Sheffield Children's Hospital, Sheffield
  - Southampton University Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency